CLINICAL TRIAL: NCT01091493
Title: Utility of Antibiotic Treatment in Acute Non-purulent Exacerbations of COPD: a Double Blinded, Randomized, Placebo-controlled Trial of Security and Efficacy
Brief Title: Antibiotic or Not in Non-purulent Exacerbations of COPD: a Trial of Security and Efficacy
Acronym: AEPOC-ATB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Nestor Soler Porcar, MD, PhD, Especialista Senior, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AEPOC-ATB
Record Dates: First submitted 2010-03-19; First posted 2010-03-24 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-Antibiotic (No Intervention): Patients will not receive antibiotics, although the study is double-blind.
- Antibiotic (Active Comparator): Patients will receive in a masked way, moxifloxacin.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Moxifloxacin — Moxifloxacin 400 mg administered once a day for 5 days
  Other Names: Actira
  Arms: Antibiotic

SUMMARY:
COPD is one of the most important causes of morbidity and mortality and supposes a sanitary problem in Europe and USA. Patients with COPD usually have 1-2 episodes of acute exacerbation of COPD (AECOPD) per year, being these the principal causes of of hospitalizations, respiratory problems and medical visits. After an episode of AECOPD, the majority of patients develop a transitory (or permanent) worsening in their quality of life and 50% of them will require a new hospitalization. Globally, a 75%& of the exacerbations might be associated with a respiratory tract infection, and among them, 50% might be related to bacteria and in 45% an evidence of viral infection could be documented. Even though the antibiotic treatment might not be useful for a majority of patients with AECOPD, is generalized its use(almost an 85% in some series) in hospitalized patients. The non-controlled use of antibiotics in AECOPD results in a very expensive disease and raises the rate of resistance of bacteria. The available literature have shown that there's a relation between exacerbations and infections, based on sputum samples.

In summary, is well known that at least a 50% of the episodes of AECOPD might be associated with pathogenic bacteria in the lower respiratory tract. Prescription of antibiotics is wide and generalized in hospitalized patients. Clinical trials have shown correlation between AECOPD with sputum purulence (which correlates with presence of bacteria), however they've not included NON-purulent AECOPD, even though they're a significative group of patients hospitalized by this cause too. It's necessary to evaluate the efficacy nor the security of antibiotic treatment in this group of patients in a well designed trial.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis according to GOLD guidelines
* Hospitalization for any acute exacerbation of chronic obstructive pulmonary disease
* Failure of outpatient treatment
* Increasing of dyspnea in the last days
* Comorbidity that causes detriment of respiratory function

Exclusion Criteria:

* Life expectancy of less than 6 months
* Mechanical Ventilation
* Cardiovascular condition that causes exacerbation
* Immunosuppression
* Pulmonary infiltrates that suggest pneumonia
* Antibiotic treatment in the last month
* Pregnancy
* ECG with a large QT segment
* Hypokalemia
* Hepatic failure or renal failure

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-07; Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment WITHOUT antibiotics in non-purulent exacerbations of COPD | Six months

SECONDARY OUTCOMES:
Efficacy/Safety in treatment on re-hospitalizations at six months. | Six monts
In-hospital stay (days) | Six months
All cause mortality | One and Six months
Quality of Life (QoL) measured by the Saint George Respiratory Questionnaire | Hospitalization day 1 and six months
  This item will be measured by the application of the Saint George Respiratory Questionnaire (SGRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Soler, MD,PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (4):
- Spain (4):
  - Hospital Miquel Servet, Zaragoza, Aragon
  - Fundacio Clinic Per la Recerca Biomèdica - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Fundació La Fe- Hospital La Fe, Valencia, Valencia
  - Hospital Clínica Platón, Barcelona

REFERENCES:
- [Background] Murray CJ, Lopez AD, Black R, Mathers CD, Shibuya K, Ezzati M, Salomon JA, Michaud CM, Walker N, Vos T. Global burden of disease 2005: call for collaborators. Lancet. 2007 Jul 14;370(9582):109-110. doi: 10.1016/S0140-6736(07)61064-2. No abstract available. PMID 17630021
- [Background] Connors AF Jr, Dawson NV, Thomas C, Harrell FE Jr, Desbiens N, Fulkerson WJ, Kussin P, Bellamy P, Goldman L, Knaus WA. Outcomes following acute exacerbation of severe chronic obstructive lung disease. The SUPPORT investigators (Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments). Am J Respir Crit Care Med. 1996 Oct;154(4 Pt 1):959-67. doi: 10.1164/ajrccm.154.4.8887592.
- [Background] Snow V, Lascher S, Mottur-Pilson C; Joint Expert Panel on COPD of the American College of Chest Physicians and the American College of Physicians-Amercian Society of Internal Medicine. The evidence base for management of acute exacerbations of COPD: clinical practice guideline, part 1. Chest. 2001 Apr;119(4):1185-9. doi: 10.1378/chest.119.4.1185. No abstract available. PMID 11296188